CLINICAL TRIAL: NCT01491152
Title: Side-alternating Whole Body Vibration in Children With Cerebral Palsy (CP) From 12 Months of Age - Pilot Study
Brief Title: Pilot Study of Whole Body Vibration for Children With Cerebral Palsy (CP) From 12 Months of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Christina Stark, Staff member at the muscle-bone research group, University of Cologne
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Uni-Koeln-1527
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2013-09

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral Palsy; Whole Body Vibration; Infant; Motor development; Physiotherapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBV Training (Experimental)
  Interventions: Device: Galileo® tilt table for children
- Control (No Intervention): No WBV Training. Standard of Care.

INTERVENTIONS:
Device: Galileo® tilt table for children — Two weeks of introduction and 12 weeks of training with side-alternating whole body vibration (WBV) (Galileo® tilt table)
  Other Names: Novotec Medical, Pforzheim, Germany
  Arms: WBV Training

SUMMARY:
Cerebral Palsy (CP) is the most common cause of physical disability in childhood. Up to day the investigators have treated children diagnosed cerebral palsy with side-alternating whole body vibration (System Galileo®) from the age of two years on. Considering verticalisation (standing and walking) at about 12 months of age in a normal developing child the investigators suggest the introduction of verticalisation with whole body vibration to a child with CP at this early age in order to enhance motor development and participation.

In this pilot study the investigators will test the feasibility and the effect on motor development of whole body vibration in children with CP from 12 months of age. The investigators will investigate the effect of whole body vibration on motor performance, independence in all day living situations, quality of life and contractures compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed CP
* ≥ 12 months and ≤ 24 months of age (prematures corrected age)
* GMFCS level II, III, IV
* Inability to stand and walk
* Written informed consent of legal guardian

Exclusion Criteria:

* Chronic infectious disease
* Epilepsy not responding to therapy
* Additional severe congenital disorder (e.g. congenital heart disorder)
* Surgery in previous three months
* Hernia requiring surgery
* Treatment with Botulinumtoxin
* Acute Thromboses
* Implants and tendinitis in body parts to be trained
* Acute inflammation in the musculoskeletal system
* Slipped disc
* Rheumatoid arthritis
* Fractures in previous three months
* Intracerebral bleeding in previous three months
* Planned surgery in study period
* Participation at another interventional trial
* Gall stones, kidney stones and pregnancy of the person who trains with the child

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change of gross motor function (GMFM-66) | Baseline (T0), week 14 (T1, after training) und week 28 (T2, after follow-up)

SECONDARY OUTCOMES:
Participation in activities in daily life (PEDI) | Baseline (T0), week 14 (T1, after training) und week 28 (T2, after follow-up)
Health-related quality of life (PedsQL) | Baseline (T0), week 14 (T1, after training) und week 28 (T2, after follow-up)
Passive Range of Motion (PROM) | Baseline (T0), week 14 (T1, after training) und week 28 (T2, after follow-up)
Training compliance | Baseline (T0), week 14 (T1, after training) und week 28 (T2, after follow-up)
  Training compliance will be evaluated by the number of completed training units during the 14-week training period at home. Each training session will be documented in the patient diary (training protocol). Additionally the Galileo® WBV system will automatically record all training sessions performed on the device as date, time and duration of training session.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Stark, MSc., Principal Investigator — Children's Hospital University of Cologne; Peter Herkenrath, Dr., Principal Investigator — Children's Hospital University of Cologne; Eckhard Schoenau, Prof., Study Chair — Children's Hospital University of Cologne
Locations (1):
- Children's Hospital University of Cologne, Cologne, Germany